CLINICAL TRIAL: NCT05800314
Title: Effectiveness of Different Scoring Systems in Prediction of Prognosis in Acute Intoxicated Cases in Assiut University Hospitals
Brief Title: Effectiveness of Different Scoring Systems
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Raghda Mostafa Shaban Ali, Effectiveness of Different Scoring Systems in Prediction of Prognosis in Acute Intoxicated Cases in Assiut University Hospitals, Assiut University
Other Study IDs: Scoring systems
Record Dates: First submitted 2023-03-02; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Assessment of the effectiveness of a validated poisoning specific scoring system (new poisoning mortality [PMS]) and other commonly used scoring systems for all acutely ill patient (Simple clinical score [SCS] and Rapid Emergency Medicine Score [REMS]) at Assiut university hospitals.
2. Comparison between these scoring systems in terms of sensitivity and specificity in both children and adults.
3. Design a toxicological sheet for Assiut poison control center that include this poisoning scoring system so it could help in assessing prognosis of acute poisoned cas

DETAILED DESCRIPTION:
Acute poisoning is a global health problem. Prevention of mortality in both intentional and accidental poisonings is essential(Cheung et al., 2018) Regarding prevalence in Egypt, 38470 pediatric patients presentedd to Ain Shams University -Poisoning Toxicology Center(ASU-PTC) 2009-2013 (Sonya et al., 2016) .Also, 937 adult poisoned patients were admitted to Tanta Emergency University hospital in 2012 (Enas, 2012).

Mortality prediction in acute poisoning cases has been explored by applying various clinical scoring systems used in critical care (Alizadeh et al, 2014; Banderas-Bravo et al., 2017) .

There are different non-specific scoring systems that depend physiological variables only such as:

1. The acute physiology and chronic health evaluation (APACHE) score
2. Simplified Acute physiology score (SAPS) They are commonly applied tools in the intensive care unit; they are used for predicting the outcomes in poisoning cases. But they became of limited utility because they are time consuming. (Bilgin et al., 2005).

There are other non-specific scoring system but non time consuming such as

1. Rapid Emergency Medicine Score (REMS) was a powerful predictor of in hospital mortality in patients attending the ED
2. Simple Clinical Score (SCS) a quickly and accurately identifying patients at both a low and high risk of death. (J Kellett,et al ,2006) New Poisoning Mortality Score (PMS):is specific scoring system that depends on demographic variables, poisoning related variables and vital signs, so accurately predicted the probability of death for patients with acute poisoning. This could contribute to the clinical decision making for patients with acute poisoning at the ED (Han et al., 2021). Results indicated that 724 poisoning cases were admitted to Children's Hospital during the year 2012 in Assuit governorate, Prediction of prognosis in patients with acute poisoning has a clinical significance i.e., it helps in timely and appropriate treatment. However, toxicology research lacks a well-accepted method for assessing the severity of poisoning (Cheung et al., 2018). There is a lack in using and including this scoring systems in daily assessing of patients. Thus, the objective of this study is to assess the efficacy of a poisoning specific scoring system (PMS) and other nonspecific, physiologic, and rapid scoring systems (REMS and SCS). This could assist in treatment and therapeutic decision making at early stages for patients with acute poisoning.

ELIGIBILITY:
Inclusion Criteria:

- 1-All symptomatic cases with acute toxicity admitted to emergency units of Assiut university hospital and Assiut University Children hospital. Diagnosis based on history taking, clinical examination of the patients, toxicological investigations if available, and exclusion of relevant differential diagnoses.

2- Willing and able to comply with the study procedures and provide a written informed consent to participate in the study

Exclusion Criteria:

* Patients with a history of renal, hepatic, CNS, and cardiac diseases and cance
* Patients who will be transferred from the initial ED to another hospital. Patients who have incomplete data on poisoning-related variables
* Pregnant women.- Patient presented with a delay more than 48

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Prospective cross- sectional study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
need for intubation, need for ICU and hospital | Baseline
  The patients need for intubation, ICU,hospital stay

SECONDARY OUTCOMES:
Mortality was assessed during the hospital stay of the patients till discharge. | Baseline
  Measure the mortality for acute poisoning

IPD SHARING:
Plan to Share IPD: Undecided